CLINICAL TRIAL: NCT03570762
Title: Long Term Outcomes Of Hybrid Percutaneous Intervention With Bioresorbable Vascular Scaffolds And Drug Eluting Stents For Complex Coronary Artery Lesions
Brief Title: Long Term Outcomes Of Hybrid Percutaneous Approach
Status: Completed | Type: Observational
Sponsor: Liv Hospital Ankara (Other)
Responsible Party: Principal Investigator, Erol Kalender, Principal investigator, Liv Hospital Ankara
Other Study IDs: 322157920101986
Record Dates: First submitted 2018-06-18; First posted 2018-06-27 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Coronary Artery Disease
Keywords: bioresorbable vascular scaffold
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: US Export: Yes

INTERVENTIONS:
Procedure: hybrid percutaneous intervention

SUMMARY:
Bioresorbable vascular scaffolds (BVS) are considered as a new revolution in coronary intervention due to their potential advantages for long term follow up. However, current generation BVS have also some drawbacks that restrict the use for complex lesions. Using BVS and drug eluting stents (DES) together -implanting DES for BVS inappropriate segments -may be a feasible option to avoid the disadvantages of permanent foreign body and to reduce very late adverse events. In this context, we investigated the clinical outcomes following treatment with hybrid strategy with concomitant use of BVS and DES for complex lesions. A single center retrospective cohort was performed enrolling 40 patients with complex lesions treated with hybrid approach from February 2015 up to April 2017. Lesion segments with a large plaque burden and/or severe calcification, aorto-ostial and bifurcation lesions that may be unfavorable for BVS, treated with DES. BVS and DES were implanted with minimal overlap of DES and BVS struts. The primary end-point was target lesion failure (TLF) which was a composite of cardiac death, target vessel myocardial infarction and target lesion revascularization (TLR). During follow-up, coronary angiography was performed when patients had ischemic symptoms.

ELIGIBILITY:
Inclusion Criteria:

* treated with BVS in combination with DES

Exclusion Criteria:

* treated with only DES or BVS

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: cardiology clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
target lesion failure | 2 year
  a composite of cardiac death, target vessel myocardial infarction and target lesion revascularization

IPD SHARING:
Plan to Share IPD: Undecided